CLINICAL TRIAL: NCT03273530
Title: Integrated Supported Employment for People With Schizophrenia in Mainland China: A Randomized Controlled Trial
Brief Title: Integrated Supported Employment in Mainland China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Professor and Department Head of Rehabilitation Sciences, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201415
Record Dates: First submitted 2017-08-24; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Integrated Supported Employment (Experimental): Individual placement support intervention plus work-related social skills training
  Interventions: Other: Integrated Supported Employment
- Individualised Placement Support (No Intervention): Individual placement support intervention with pre-vocational training followed by placing individual participants to the job according to their preference and abilities
- Traditional Vocational Rehabilitation (No Intervention): general pre-vocational training and placement

INTERVENTIONS:
Other: Integrated Supported Employment — vocational assessment followed by job placement and on-going work-related social skills revision and reinforcement
  Arms: Integrated Supported Employment

SUMMARY:
In this randomized controlled trial, the researchers investigated the effectiveness of integrated supported employment (ISE) as compared with individual placement and support (IPS) and traditional vocational rehabilitation (TVR) for people with schizophrenia in mainland China.

DETAILED DESCRIPTION:
One hundred and sixty-two participants with schizophrenia were randomly assigned to ISE (n = 54), IPS (n = 54), and or TVR (n = 54). Blinded assessments of employment status, job tenure, and psychological outcomes were conducted at admission, completion of the 3-mo program, and follow-up at 7, 11, and 15 mo.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Diagnosis of schizophrenia for at least 2 years
* Being unemployed
* Willing to give informed consent
* Having no obvious cognitive, learning, or neurological impairment
* Having completed primary school education
* Having a desire to work

Exclusion Criteria:

• Having score lower than 18 on the 30-item Mini-Mental State Examination

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2015-08-15 (Actual); Study Completion 2015-12-20 (Actual)

PRIMARY OUTCOMES:
Employment rate | 4 months
  employment status, employed or unemployed

SECONDARY OUTCOMES:
Job tenure, duration | completion of the 3-mo program, and follow-up at 7, 11, and 15 mo.
  how long the job lasts

CONTACTS AND LOCATIONS:
Overall Officials: Hector WH Tsang, PhD, Principal Investigator — HKPolyU

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided

REFERENCES:
- [Derived] Zhang GF, Tsui CM, Lu AJB, Yu LB, Tsang HWH, Li D. Integrated Supported Employment for People With Schizophrenia in Mainland China: A Randomized Controlled Trial. Am J Occup Ther. 2017 Nov/Dec;71(6):7106165020p1-7106165020p8. doi: 10.5014/ajot.2017.024802. PMID 29135426